CLINICAL TRIAL: NCT01315873
Title: Phase II Trial of Bortezomib and Bendamustine in the Treatment of Relapsed/Refractory Myeloma
Brief Title: Bortezomib and Bendamustine to Treat Relapsed/Refractory Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left the institution before all data analysis was completed
Sponsor: NYU Langone Health (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-02009
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Multiple Myeloma
Keywords: myeloma; multiple myeloma; relapsed myeloma; refractory myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bendamustine Hydrochloride; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bortezomib and Bendamustine (Experimental)
  Interventions: Drug: Bendamustine; Drug: Bortezomib

INTERVENTIONS:
Drug: Bendamustine — On days 1 and 4 of each cycle, bendamustine is given at 90 mg/m^2 after bortezomib . Patients will be dose reduced to 75 mg/m^2, and then to 60 mg/m^2 bendamustine on days 1 and 4 if ANC is not >1 x 10^9/L and platelets are not >50 x 10^9/L on day 1 of each cycle.
  Patients will be treated until disease progression after at least one cycle of treatment.
  Other Names: Bendamustine HCl; Treanda
Drug: Bortezomib — On days 1 and 4 of each cycle, bortezomib is given first at 1.3 mg/m^2 followed by bendamustine given at 90 mg/m^2. Patients will be dose reduced to 75 mg/m^2, and then to 60 mg/m^2 bendamustine on days 1 and 4 if ANC is not >1 x 10^9/L and platelets are not >50 x 10^9/L on day 1 of each cycle.
  Patients will be treated until disease progression after at least one cycle of treatment.
  Other Names: Velcade

SUMMARY:
Patients with myeloma that has either not responded to previous treatment or has returned after previous treatment will be given a combination of the drugs bendamustine and bortezomib.

The bortezomib and bendamustine will be given using an intravenous line (IV) on days 1 and 4 of each cycle, with bortezomib being given first, before each dose of bendamustine. Each cycle will be 28 days long, so patients will be treated the first week of each cycle and then have 3 weeks 'off' (without any treatment). Disease assessments will be performed on day 22 of each cycle. Patients will receive the study drugs until their disease progresses or they are withdrawn from the study.

In other studies, bendamustine seems to work well with other drugs. Thus, this study hopes to show that the combination of bortezomib and bendamustine will have activity in relapsed/refractory myeloma.

DETAILED DESCRIPTION:
Patients with relapsed and refractory myeloma who have a measurable paraprotein in the serum or urine or measurable protein by Freelite or measurable disease by plasmacytoma will be given a combination of bendamustine and bortezomib each cycle. Response rate (PR or better after 2 cycles) and duration of response will be assessed. Therapy will be continued until disease progression. The bendamustine would be used in a day 1, day 4 dosing schedule after each dose of bortezomib to take advantage of the chemosensitizing properties of bortezomib. This minimizes the days of treatment to just the first week and allows rebound of blood counts. This will be a phase II trial with dose reduction as necessary.

Bendamustine is a drug which appears to be non-cross-resistant with other alkylating agents in vitro and in vivo. Thus, we hypothesize that the combination of bortezomib and bendamustine will have activity in relapsed/refractory myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent
2. Age 18 years or older
3. Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
4. Male subject agrees to use an acceptable method for contraception for the duration of the study.
5. Diagnosis of multiple myeloma based on standard criteria as follows:

   Major Criteria
   * Plasmacytomas on tissue biopsy
   * Bone marrow plasmacytosis (>30% plasma cells)
   * Monoclonal immunoglobulin spike on serum electrophoresis (IgG >3.5 g/dL or IgA >2.0 g/dL) or kappa or lambda light chain excretion >1 g/day on 24 hour urine protein electrophoresis

   Minor Criteria
   * Bone marrow plasmacytosis (10 to 30% plasma cells)
   * Monoclonal immunoglobulin present but of lesser magnitude than given under major criteria
   * Lytic bone lesions
   * Normal IgM <50 mg/dL, IgA <100 mg/dL, or IgG <600 mg/dL
   * Any of the following sets of criteria will confirm the diagnosis of Multiple Myeloma:

     * Any two of the major criteria or
     * 1 major plus 2 minor criteria.
6. Measurable disease, defined as a monoclonal immunoglobulin spike (M-Spike) on serum electrophoresis of ≥1 g/dL and/or urine monoclonal immunoglobulin spike of ≥200 mg/24 hours. Non-secretors must have measurable protein by Freelite or measurable disease by plasmacytoma to be eligible.
7. Patients must have refractory myeloma as defined by a greater than 25% increase in their M-protein. They should have progressed on bortezomib.
8. Karnofsky performance status ≥50
9. Patients treated with local radiotherapy with or without a brief exposure to steroids are eligible. Patients who require radiotherapy should have entry to the protocol deferred until the radiotherapy is completed by at least 4 weeks prior to initiation of study drug.
10. Meets the following pretreatment laboratory criteria at baseline (Day 1 of Cycle 1, before study drug administration)

    * Absolute neutrophil count ≥1 x 10^3/uL
    * Platelet count ≥75 x 10^3/uL
    * Hemoglobin ≥8.0 g/dL
    * Calculated or measured CrCL ≥ 40 mL/min
    * AST or ALT and total bilirubin < 3 x ULN
11. Echocardiogram with a >50% Ejection Fraction

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be registered on study:

1. POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M-protein) and skin changes)
2. Plasma cell leukemia
3. Receiving steroids daily for other medical conditions, e.g., asthma, systemic lupus erythematosis, rheumatoid arthritis
4. Infection not controlled by antibiotics
5. HIV infection. Patients should provide consent for HIV testing according to the institution's standard practice.
6. Known active hepatitis B or C
7. New York Hospital Association (NYHA) Class III or IV heart failure, Echo or MUGA ejection fraction < 40% (if known), or EKG evidence of acute ischemic disease
8. Other serious medical or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol
9. Second malignancy requiring treatment in the last 3 years
10. Patient has a calculated or measured creatinine clearance of <40 mL/min within 14 days before enrollment
11. Patient has >Grade 2 peripheral neuropathy within 14 days before enrollment
12. Patient has hypersensitivity to bortezomib, boron or mannitol and bendamustine
13. Positive pregnancy test in women of childbearing potential or subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum betaa human chorionic gonadotropin test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
14. Patient has received other investigational drugs with 14 days before enrollment
15. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
16. Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09; Primary Completion 2014-02 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amitabha Mazumder, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bortezomib and Bendamustine: Bendamustine: On days 1 and 4 of each cycle, bendamustine is given at 90 mg/m^2 after bortezomib . Patients will be dose reduced to 75 mg/m^2, and then to 60 mg/m^2 bendamustine on days 1 and 4 if ANC is not >1 x 10^9/L and platelets are not >50 x 10^9/L on day 1 of each cycle.
  Patients will be treated until disease progression after at least one cycle of treatment.
  Bortezomib: On days 1 and 4 of each cycle, bortezomib is given first at 1.3 mg/m^2 followed by bendamustine given at 90 mg/m^2. Patients will be dose reduced to 75 mg/m^2, and then to 60 mg/m^2 bendamustine on days 1 and 4 if ANC is not >1 x 10^9/L and platelets are not >50 x 10^9/L on day 1 of each cycle.
  Patients will be treated until disease progression after at least one cycle of treatment.
Period: Overall Study
Arm/Group | Bortezomib and Bendamustine
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib and Bendamustine
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Percent Change Response Rate (Partial Response or Better After 2 Cycles) Following Treatment With Bortezomib and Bendamustine
Description: These criteria included measures of alteration in the natural history of disease, hematologic improvement, cytogenetic response, and improvement in health-related quality of life.The IWG criteria define 4 aspects of responses based on treatment goals: (1) altering the natural history of the disease, (2) cytogenetic response, (3) hematologic improvement (HI), and (4)Quality of Life (QOL)
Time Frame: 8 weeks
Population: Participant data was not analyzed because PI left institution
Arm/Group | Bortezomib and Bendamustine
Number analyzed (Participants) | 0

2. Secondary Outcome: Toxicity of This Regimen.
Description: Study toxicity will be measured on an ongoing basis, no less then once per 28-day cycle.
Time Frame: Every 4 weeks.
Population: Participant data was not analyzed because PI left institution. Data were not available for analysis.
Arm/Group | Bortezomib and Bendamustine
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Response of This Regimen.
Description: Time from response to relapse. Response would have been assessed using European Group for Blood and Marrow Transplantation (EBMT) criteria modified to include near complete remission (nCR) and very good partial remission (VGPR
Time Frame: from initial response to relapse, up to 100 weeks.
Population: Participant data was not analyzed because PI left institution
Arm/Group | Bortezomib and Bendamustine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 8 Weeks
Arm/Group | Bortezomib and Bendamustine
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No